CLINICAL TRIAL: NCT06912477
Title: Systematic Evaluation of Endothelial Dysfunction as a Prognostic Marker for Outcomes in Women With Preeclampsia
Brief Title: Endothelial Dysfunction for Prognosis In Patients With preeClampSia
Acronym: EPICS
Status: Recruiting | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Anna Scholz, Dr. med. Anna Scholz, Heidelberg University
Other Study IDs: S-457/2024
Record Dates: First submitted 2025-03-25; First posted 2025-04-04 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Preeclampsia (PE); Hypertensive Disorder of Pregnancy
Keywords: preeclampsia; hyperspectral imaging; endothelial dysfunction
MeSH Terms: conditions — Pre-Eclampsia; Toxemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Preeclampsia: patients with diagnosis of preeclampsia according to definitions by the International Society for the Study of Hypertension in Pregnancy (n=110)
  Interventions: Diagnostic Test: Hyperspectral imaging; Diagnostic Test: Further markers of endothelial dysfunction
- Pregnancy induced Hypertension and chronic Hypertension: patients with hypertension in pregnancy without fulfilling criteria of preeclampsia (n=110)
  Interventions: Diagnostic Test: Hyperspectral imaging; Diagnostic Test: Further markers of endothelial dysfunction
- Normotensive pregnant control group: normotensive pregnancies (n=110)
  Interventions: Diagnostic Test: Hyperspectral imaging; Diagnostic Test: Further markers of endothelial dysfunction
- Non-pregnant control group: normotensive, non-pregnant women (n=55)
  Interventions: Diagnostic Test: Hyperspectral imaging; Diagnostic Test: Further markers of endothelial dysfunction

INTERVENTIONS:
Diagnostic Test: Hyperspectral imaging — Hyperspectral imaging will be performed at study inclusion and will be repeated longitudinally every 1-2 days until delivery and on the first and second day after delivery. After a baseline measurement, a blood pressure cuff is inflated on the upper arm to 50 mmHg above the systolic blood pressure for 5 minutes, and then the hyperspectral imaging measurement is repeated.
  Blood samples are collected at study inclusion and on the first and second day after delivery and are processed within the Department of Gynecology and Obstetrics of the Heidelberg University Hospital.
Diagnostic Test: Further markers of endothelial dysfunction — At study inclusion: 1. blood samples will be collected for the measurement of EASIX and cardiac/endothelial markers; 2. sublingual in vivo microscopy will be performed (requires about 20 minutes and can be compared to a sublingual temperature measurement); 3. Doppler ultrasound will be performed to evaluate uterine and ophthalmic arteries.
  Blood samples will also be collected at the first and second day after delivery.

SUMMARY:
Preeclampsia is a pregnancy-specific hypertensive disorder and can progress rapidly to severe adverse outcomes affecting both the mother and the fetus. Endothelial and microcirculatory dysfunction mediate systemic preeclampsia-related organ dysfunctions. Changes in endothelial and vascular function in preeclampsia have been demonstrated through reduced flow-mediated vasodilation as a result of reduced availability of nitric oxide, which potentially persists up to several years postpartum. Hyperspectral imaging is a new innovative technology that allows to assess the peripheral microcirculation and perfusion non-invasively and contactless, but has never been evaluated in the context of preeclampsia before.

This EPICS project (Endothelial dysfunction for Prognosis In patients with preeClampSia) is a prospective observational study and aims to investigate hyperspectral imaging as a new potential diagnostic and prognostic marker in preeclampsia.

DETAILED DESCRIPTION:
Preeclampsia is defined as hypertension combined with features of multi-organ dysfunction and can progress rapidly to severe adverse outcomes affecting both the mother and the fetus. Endothelial dysfunction is a key driver in the pathophysiology of preeclampsia mediating the systemic complications of this multi-organ disease. Changes in endothelial and vascular function in preeclampsia have been observed through reduced flow-mediated vasodilation, which occurs due to diminished nitric oxide availability and may persist for years after childbirth. Although symptoms of preeclampsia often resolve spontaneously after delivery, affected women will face a significantly increased risk of long-term cardiovascular complications. Thus, preeclampsia is viewed as an individual female-specific cardiovascular risk factor.

Beyond this background, hyperspectral imaging as an assessment of peripheral microcirculation and tissue perfusion appears to be a suitable method. Hyperspectral imaging is an innovative technique that visualizes hemodynamic changes by displaying the oxygen saturation of hemoglobin in the capillary system, the distribution of hemoglobin in the tissue, and the relative tissue water content. Hyperspectral imaging has not yet been studied in obstetrics or in the context of preeclampsia before. Given the well-documented microcirculatory disturbances associated with preeclampsia, the investigators hypothesize hyperspectral analysis as a valuable tool to bridge a diagnostic gap that might be useful to tailor individualized obstetric care of patients with preeclampsia.

Recently the "Endothelial Activation and Stress Index" (EASIX) was evaluated as prognostic marker in preeclampsia by the investigator group. EASIX is based on lactate dehydrogenase, platelets, and creatinine and was originally developed as simple score to predict endothelial-related complications after allogenic stem cell transplantation. However, the exact relationship of EASIX to endothelial cell biology and microcirculation requires further clarification. The investigators hypothesize that a reduced peripheral microcirculation will mediate direct interactions of platelets with endothelial cells, resulting in cellular damage (increased LDH), loss of platelets due to activation and microembolism, and lead to kidney damage.

The EPICS study (Endothelial dysfunction for Prognosis In patients with preeClampSia) is the first prospective study to investigate hyperspectral imaging in women with preeclampsia. The aim of this study is to evaluate whether and how changes in microcirculation in women with preeclampsia can be detected with hyperspectral imaging compared to women with pregnancy-induced hypertension, normotensive pregnant women and non-pregnant controls and whether microcirculatory perfusion quality is associated with other biochemical markers such as EASIX or markers of endothelial dysfunction. Furthermore, the EPICS study aims to evaluate the predictive performance of hyperspectral imaging with or without combination of other biochemical markers for adverse maternal and perinatal outcomes and the remaining time until delivery in patients with preeclampsia.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancies
* Age ≥ 18 years
* Patient's ability to provide consent
* written informed consent

Exclusion Criteria:

* Lack of consent
* Language barrier
* Dark to very dark skin type
* Severe fetal chromosomal/genetic/structural anomalies
* Laboratory changes in LDH, creatinine, or platelets due to other causes (e.g., isolated thrombocytopenia, e.g., immune thrombocytopenia, carcinoma)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are admitted to the Department of obstetrics at Heidelberg University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Time Until Delivery | observation period until 6 months after delivery
  Time period between date of study inclusion (diagnostic tests) to delivery

SECONDARY OUTCOMES:
maternal adverse event | observation period until 6 months after delivery
  composite adverse maternal outcome (categorical, yes/no): death, acute kidney injury, cardiorespiratory complication (e.g. pulmonary edema), eclampsia, cerebrovascular event, hematological complication, hepatic complication, postpartum hemorrhage, the Hemolysis, Elevated Liver enzymes, Low Platelets (HELLP) syndrome, placental abruption
perinatal adverse event | observation period until 6 months after delivery
  composite perinatal endpoint (categorical, yes/no): neonatal mortality, stillbirth, preeclampsia-related preterm delivery, respiratory distress syndrome, neonatal seizures, intraventricular hemorrhage, necrotizing enterocolitis, birthweight <10th percentile, admission to neonatal unit, respiratory support
maternal cardiovascular outcome: persistence of hypertension | observation period until 6 months after delivery
  number of participants with persisting hypertension
maternal cardiovascular outcome: blood pressure | observation period until 6 months after delivery
  blood pressure (mmHg)
maternal cardiovascular outcome: antihypertensive medication | observation period until 6 months after delivery
  number of participants who required antihypertensive medication initiation or dose adjustment
maternal cardiovascular outcome: readmission | observation period until 6 months after delivery
  number of participants who required readmission for hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Dr. med. Alexandra von Au, Principal Investigator — University Heidelberg
Locations (1):
- Heidelberg University Hospital, Department of Gynecology and Obstetrics, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided